CLINICAL TRIAL: NCT06697483
Title: Risk Stratification and MRD-driven Maintenance for Multiple Myeloma After Autologous Stem Cell Transplantation
Brief Title: Risk Stratification and MRD-driven Maintenance for MM After ASCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jin Lu, MD, Principal of Investigator, Peking University People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024PHB165-001-20240930
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Multiple Myeloma
Keywords: R2-ISS stage; Minimal Residual Disease; Lenalidomide; Daratumumab
MeSH Terms: conditions — Multiple Myeloma; Neoplasm, Residual | interventions — daratumumab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lenalidomide (Other): For patients with low-risk or intermediate-low risk and minimal residual disease negativity before maintenance
  Interventions: Drug: Lenalidomide
- Daratumumab and Lenalidomide (Other): For patients with high-risk or intermediate-high risk OR minimal residual disease posivitity before maintenance
  Interventions: Drug: Daratumumab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Daratumumab — Patients who are R2-ISS 3 or 4 OR MRD (Minimal Residual Disease) positivity will receive daratumumab plus lenalidomide maintenance.
  Arms: Daratumumab and Lenalidomide
Drug: Lenalidomide — Patients are R2-ISS 1,2 and MRD (Minimal Residual Disease) negative after autologous stem cell transplantation.
  Patients will receive the single drug lenalidomide maintenance.

SUMMARY:
This study evaluates the maintenance strategy based on risk stratification and MRD status after stem cell transplantation.

This is a single-arm, multicenter, prospective study. Participants who are R2-ISS 1,2 and MRD negative receive the single drug lenalidomide maintenance. In other circumstances, for example, patients who are R2-ISS 3 or 4 will receive daratumumab combined with lenalidomide regardless of MRD status, while patients with MRD positivity will also receive daratumumab plus lenalidomide maintenance.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed multiple myeloma with a history of a minimum of 4 cycles of induction therapy, have received high-dose therapy (HDT) and autologous stem cell transplantation (ASCT) within 12 months of the start of induction therapy, and be within 6 months of ASCT.
2. Must have a partial response (PR) or better response before maintenance.
3. Must have an Eastern Cooperative Oncology Group performance status score of 0, 1, or 2.
4. This study allows for post-ASCT consolidation therapy.
5. ANC ≥ 1.0 x 10^9/L, Hb ≥ 85 g/L PLT ≥ 75 x 10^9/L (if BMPC < 50%) or PLT ≥ 50 x 10^9/L (if BMPC ≥ 50%).
6. No active infection.
7. a).TBIL<1.5 x upper limit of normal (ULN) (<3 x ULN in patients with Gilbert's syndrome); b).AST and ALT <3 x ULN.; c. Creatinine clearance ≥ 45mL/min.

Exclusion Criteria:

1. Must not refractory or non-tolerate to lenalidomide in Arm A.
2. Must not refractory or non-tolerate to lenalidomide and daratumumab in Arm B.
3. Must not have progressed on multiple myeloma (MM) therapy before screening
4. Chronic obstructive pulmonary disease (COPD) with FEV1 less than 50 % of predicted normal；
5. Have known moderate or severe persistent asthma within the past 2 years or current uncontrolled asthma of any classification
6. History of stroke or serious thrombotic event within 12 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
MRD (Minimal Residual Disease) status at 12 months after maintenance | 12 months
  Bone marrow minimal residual disease status at 12 months after maintenance

SECONDARY OUTCOMES:
CR+VGPR | 12 months
  complete response plus very good partial response at 12 months from maintenance
Estimated 3 year-PFS | 3 years
  Estimated 3 year progression free survival
Estimated 3 year OS | 3 years
  Estimated 3 year overall survival
TRAEs | 3 years
  Treatment related adverse events

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Fuxing Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang

IPD SHARING:
Plan to Share IPD: No